CLINICAL TRIAL: NCT02596295
Title: Human Milk Sample Collection From Israeli Mothers and Its Analysis and Correlation Between Composition, Demographics and Diet
Brief Title: Human Milk Sample Composition in Israeli Mothers and Correlation With Their Diet
Status: Completed | Type: Observational
Sponsor: Enzymotec (Industry)
Responsible Party: Sponsor
Other Study IDs: HM001
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Breast Milk Collection
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mothers for term infants: Lactating mothers
- Mothers for preterm infants: Lactating mothers

SUMMARY:
The study will collect human milk from 100 mother of term infants 2-3m after delivery and from 50 mothers of preterm infants 14 and 30 days after delivery. Sample content will be analysed and statistical analysis will look at correlation between demographics, dietary habits and milk composition.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy mothers who give birth to a healthy term infant (37-42 weeks) Mothers who intend to breastfeed the infant at least 80% of the daily feeding Mothers who can comply with the study requirements Mothers who sign the informed consent form in writing and can read and write Hebrew.

Exclusion Criteria:

* Participation in any other studies involving investigational or marketed products Is consuming alcoholic drinks and is a drug abuser. Is suffering from chronic disease Presence of psychosis and severe post-partum depression. Mothers who have given birth to twins or multiples Mothers who received chemotherapy or isotopes during pregnancy investigator's uncertainty about the willingness or ability of the mothers to understand and comply with the protocol requirements.

Infants:

Any congenital abnormality, chromosomal disorder or severe disease which could interfere with the study conduct and assessment.

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: General healthy lactating mothers
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Analysis of natural lipids in human breast milk of Israeli's mothers | 30-60 days after delivery
  exploratory study

SECONDARY OUTCOMES:
Maternal diet survey | 30-60 days after delivery
  exsploratory study

CONTACTS AND LOCATIONS:
Overall Officials: Yael Lifshitz, PhD, Study Director — Employee
Locations (1):
- Meir Hospital, Kfar Saba, State, Israel